CLINICAL TRIAL: NCT01995929
Title: Transnasal Endoscopic Evaluation of Swallowing: Functional Esophagoscopy Using an Ultrathin Video Endoscope in Neurogenic Dysphagia
Brief Title: Functional Endoscopy in Neurogenic Dysphagia
Status: Completed | Type: Observational
Sponsor: University Hospital Muenster (Other)
Responsible Party: Principal Investigator, Dr. Dirk Domagk, Prof. Dr. med. Dirk Domagk, University Hospital Muenster
Other Study IDs: 2012_2013_003; TNE_2010 (Other: University Hospital of Muenster)
Record Dates: First submitted 2013-11-18; First posted 2013-11-27 (Estimated); Last update posted 2022-11-09 (Actual); Status verified 2020-12

CONDITIONS: Neurogenic Dysphagia
Keywords: neurogenic dysphagia; transnasal endoscopy; functional endoscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- neurogenic dysphagia: Patients suffering from neurogenic dysphagia due to several reasons (e.g. Parkinson´s disease).
  Interventions: Procedure: transnasal functional endoscopy

INTERVENTIONS:
Procedure: transnasal functional endoscopy
  Other Names: ultrathin video endoscope with an outer diameter of 3.8 mm (BF-3C160, Olympus Europe)

SUMMARY:
The esophago-gastro-duodenoscopy is an endoscopic examination technique of the upper GI-tract which was founded by the German surgeon Johann Freiherr von Mikuliicz-Radecki at the end of 19th century. By this means, the luminal site of the esophagus, stomach and duodenum may be visualized after inserting a flexible endoscope through the mouth (transoral access). By the rapid technical development in the last years smaller flexible video endoscopes have been developed allowing also an alternative access to the upper GI-tract via the nose (transnasal access).

Patients with dysphagia are referred to physicians of different disciplines (gastroenterology, surgery, ear, nose, and throat (ENT) medicine, radiology, neurology) performing a variety of endoscopic and non-endoscopic techniques. Mostly, the endoscopic examination of the esophagus is done in sedated patients in left lateral examination. Typical findings during esophagoscopy might be tumors, strictures, achalasia or diverticula.

Patients suffering from neurogenic dysphagia often get caught in the trap: they find themselves somewhere in the space between gastroenterologist, neurologist, ENT-specialist and radiologist. This dilemma might be due to a lack of pathophysiological knowledge among many physicians and an inability to directly visualize the esophageal phase of deglutition. In sedated patients lying in left lateral position, endoscopists may receive a very limited impression of the function of the different phases of swallowing since this endoscopic access is a rather static one.

The focus of our observational study are patients with suspected neurogenic dysphagia. These patients shall be examined by transnasal endoscopy applying an ultrathin video endoscope with an outer diameter of 3.8 mm (BF-3C160, Olympus Europe). Patients are examined in sitting position while ingesting water and food of different consistencies (functional endoscopy). Diagnostic shall be completed and correlated by videofluoroscopy, high-resolution manometry and assessment of the clinical signs. Beside feasibility and safety as primary endpoints, secondary endpoints shall be the assessment of pathologic endoscopic findings in patients suffering from neurogenic dysphagia. The study is approved by the local Ethics Committee (AZ 2010-214-f-S).

DETAILED DESCRIPTION:
The esophago-gastro-duodenoscopy is an endoscopic examination technique of the upper GI-tract which was founded by the German surgeon Johann Freiherr von Mikuliicz-Radecki at the end of 19th century. By this means, the luminal site of the esophagus, stomach and duodenum may be visualized after inserting a flexible endoscope through the mouth (transoral access). By the rapid technical development in the last years smaller flexible video endoscopes have been developed allowing also an alternative access to the upper GI-tract via the nose (transnasal access).

Patients with dysphagia are referred to physicians of different disciplines (gastroenterology, surgery, ear, nose, and throat (ENT) medicine, radiology, neurology) performing a variety of endoscopic and non-endoscopic techniques. Mostly, the endoscopic examination of the esophagus is done in sedated patients in left lateral examination. Typical findings during esophagoscopy might be tumors, strictures, achalasia or diverticula. In sedated patients lying in left lateral position, endoscopists may, therefore, receive a very limited impression of the actual function of the different phases of swallowing since this endoscopic approach is a rather static one.

Patients suffering from neurogenic dysphagia often get caught in the trap: they find themselves somewhere in the space between gastroenterologist, neurologist, ENT-specialist and radiologist. This dilemma might be due to a lack of pathophysiological knowledge among many physicians and an inability to directly visualize the esophageal phase of deglutition.

The focus of our observational study are patients with suspected neurogenic dysphagia. These patients shall be examined by transnasal endoscopy applying an ultrathin video endoscope with an outer diameter of 3.8 mm (BF-3C160, Olympus Europe). Patients are examined in sitting position while ingesting water and food of different consistencies (functional endoscopy). Diagnostic shall be completed and correlated by videofluoroscopy, high-resolution manometry and assessment of the clinical signs. Beside feasibility and safety as primary endpoints, secondary endpoints shall be the assessment of pathologic endoscopic findings in patients suffering from neurogenic dysphagia. The study is approved by the local Ethics Committee (AZ 2010-214-f-S).

ELIGIBILITY:
Inclusion Criteria:

* patients with suspected neurogenic dysphagia, not fulfilling the exclusion criteria

Exclusion Criteria:

* Age under 18 years
* Inability to understand information for participation
* Refusal of participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The focus of our observational study are patients with suspected neurogenic dysphagia.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
Number of patients in which the procedure may be successfully performed (feasibility) | 30 minutes
  Feasibility, safety, and tolerability of the procedure

SECONDARY OUTCOMES:
Pathologic endoscopic findings in patients suffering from neurogenic dysphagia | 30 minutes
  Acquisition of pathologenic mechanism during swallowing
Number of patients with adverse events as a measure of safety and tolerability | 1 week
  safety of transnasal functional endoscopy in diagnostics of neurogenic dysphagia

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Josephs Hospital Warendorf, Warendorf, North Rhine-Westphalia
  - University Hospital of Muenster, Münster

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cheung J, Bailey R, Veldhuyzen van Zanten S, McLean R, Fedorak RN, Morse J, Millan M, Guzowski T, Goodman KJ; CANHelp working group. Early experience with unsedated ultrathin 4.9 mm transnasal gastroscopy: a pilot study. Can J Gastroenterol. 2008 Nov;22(11):917-22. doi: 10.1155/2008/323027. PMID 19018337
- [Background] Wiegand N, Bauerfeind P, Delco F, Fried M, Wildi SM. Endoscopic position control of nasoenteral feeding tubes by transnasal re-endoscopy: a prospective study in intensive care patients. Am J Gastroenterol. 2009 May;104(5):1271-6. doi: 10.1038/ajg.2009.26. Epub 2009 Mar 24. PMID 19319127
- [Background] Zhihui T, Wenkui Y, Weiqin L, Zhiming W, Xianghong Y, Ning L, Jieshou L. A randomised clinical trial of transnasal endoscopy versus fluoroscopy for the placement of nasojejunal feeding tubes in patients with severe acute pancreatitis. Postgrad Med J. 2009 Feb;85(1000):59-63. doi: 10.1136/pgmj.2008.070326. PMID 19329697
- [Background] Warnecke T, Teismann I, Oelenberg S, Hamacher C, Ringelstein EB, Schabitz WR, Dziewas R. Towards a basic endoscopic evaluation of swallowing in acute stroke - identification of salient findings by the inexperienced examiner. BMC Med Educ. 2009 Mar 10;9:13. doi: 10.1186/1472-6920-9-13. PMID 19284543
- [Background] Warnecke T, Teismann I, Oelenberg S, Hamacher C, Ringelstein EB, Schabitz WR, Dziewas R. The safety of fiberoptic endoscopic evaluation of swallowing in acute stroke patients. Stroke. 2009 Feb;40(2):482-6. doi: 10.1161/STROKEAHA.108.520775. Epub 2008 Dec 12. PMID 19074481
- [Background] Warnecke T, Teismann I, Zimmermann J, Oelenberg S, Ringelstein EB, Dziewas R. Fiberoptic endoscopic evaluation of swallowing with simultaneous Tensilon application in diagnosis and therapy of myasthenia gravis. J Neurol. 2008 Feb;255(2):224-30. doi: 10.1007/s00415-008-0664-6. Epub 2008 Jan 28. PMID 18217186
- [Background] Herrmann IF, Scarpignato C. [Functional endoscopy : the physiological and pathophysiological basis of reflux disease, diagnosis and therapy]. HNO. 2009 Dec;57(12):1221-36. doi: 10.1007/s00106-009-1934-z. German. PMID 19924362
- [Derived] Ruckert J, Lenz P, Heinzow H, Wessling J, Warnecke T, Herrmann IF, Strahl M, Lenze F, Nowacki T, Domagk D. Functional endoscopy in neurogenic dysphagia: a feasibility study focusing on the esophageal phase of swallowing. Endosc Int Open. 2021 Apr;9(4):E646-E652. doi: 10.1055/a-1380-3224. Epub 2021 Apr 15. PMID 33880400